CLINICAL TRIAL: NCT05399823
Title: The Effect of Taping in Addition to Self-stretching Exercise on Thoracic Kyphosis Angle, Neck Pain and Quality of Life in Elderly People With Hyperkyphosis
Brief Title: The Effect of Taping in Addition to Self-stretching Exercise in the Elderly People With Hyperkyphosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özge Gökalp, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/0111
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Physical Performance
Keywords: Exercise; Kinesiotape; Kyphosis; Elderly
MeSH Terms: conditions — Motor Activity; Kyphosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self Stretching and Kinesio Taping Group (Experimental): Kinesio taping in addition to self stretching exercises will be given for 15-20 minutes at home or in the office every day for four weeks.
  Interventions: Other: Exercise
- Self Stretching and Sham Taping Group (Sham Comparator): Sham kinesio taping in addition to self stretching exercises will be given for 15-20 minutes at home or in the office every day for four weeks.
  Interventions: Other: Exercise
- Self Stretching Group (Active Comparator): A program consisting of stretching exercises for pectoral, erector spinae, latismus dorsi, multifidus, rhomboid and trapezius muscles will be given for 15-20 minutes at home or in the office every day for four weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Strecthing exercises will given for 15-20 minutes everyday for four weeks

SUMMARY:
Aim: The aim of the study is to investigate the effectiveness of kinesio taping and sham taping in addition to self-stretching exercise on hyperkyphosis angle, neck pain and quality of life in elderly individuals with hyperkyphosis.

Method: 60 elderly individuals with hyperkyphosis aged 60-85 years will be included in the study. Subjects will be divided inti three groups. Kinesio taping, sham taping and self-stretching exercise. The kinesio taping group will be given kinesio taping in addition to self stretching exercises. The second sham taping group will be given sham kinesio taping in addition to self stretching exercises. The third self-stretching group will be given a program consisting of stretching exercises for pectoral, erector spinae, latismus dorsi, multifidus, rhomboid and trapezius muscles. Individuals will be asked to do these exercises on their own for 15-20 minutes at home or in the office every day for four weeks. Before and after the study, the subjects will be test for the kyphosis angle will be evaluated with a flexible ruler and Scoliosis Research Society Outcome questionnaire (SRS22) will be used to evaluate spinal curvatures.The Neck Disability Questionnaire will be used to evaluate neck pain. The occiput-neck distance and mini mental test will be used in this srudy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer female and male individuals between the aged of 60-85 years,
* Kyphosis angle is greater than 56 degrees in women and 62 degrees in men,
* Individuals who have not physiotherapy in the last 6 months,
* Individuals who have not phsical activity in the last 6 months.

Exclusion Criteria:

* Individuals with any thoracic scoliosis and Scheuermann's disease,
* Individuals who having a kinesio tape allergy or developing an allergy while working.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-08-28 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in the kyphosis angle to be evaluated by a flexible ruler | Baseline and at the end of 4 weeks
  C7 and T12 vertebrae will be taken as reference in the measurement of the kyphosis angle. The Q angle is calculated by measuring the distances between the points taken as criteria.

SECONDARY OUTCOMES:
Chane in the spinal curvature to be evaluated by Scoliosis Research Society Outcome Questionnaire (SRS22) | Baseline and at the end of 4 weeks
  The SRS-22 scale is a scale developed by the Scoliosis Research Society to evaluate all spinal curvatures. The scale consists of 22 questions and five subgroups. Subgroups; pain, body image, spine functions, mental health and satisfaction with treatment. Scores are calculated by assigning an answer value to all 22 questions within a five-point indicator chart.

OTHER OUTCOMES:
Change in the level of neck pain and neck dysfunction to be evaluated by Neck Disability Questionnaire | Baseline and at the end of 4 weeks
  It is a patient-filled, condition-specific functional status questionnaire consisting of 10 items including pain, self-care, lifting, reading, headache, concentration, work, driving, sleep, and recreation. Each section is scored on a scoring scale from 0 to 5; where zero means 'No Pain' and 5 means 'Worst pain imaginable'.
Change in the level of neck disability to be evaluated by Occiput-Wall Distance test | Baseline and at the end of 4 weeks
  For the measurement of occiput-wall distance, the patient stands in a standing position with his back to the wall with his hips and knees as straight as possible and tries to touch his head to the wall as much as possible in a neutral position. At this time, the occiput wall distance is measured in cm. The test is repeated 3 times and the mean distance is used to divide the participants into 3 groups according to the severity of kyphosis, including mild (≤5.0 cm), moderate (5.1-8.0 cm), and severe (> 8.0 cm).
Cognitive level of the subjects to be evaluated by Standardized Mini Mental Test | Baseline
  Different cognitive abilities such as orientation, long and short term memory, attention, calculation, motor function and perception, remembering, language, and visuospatial abilities are used between 24-30 points normal, 18-23 points mild dementia, 17 points and below severe dementia it is compatible.

CONTACTS AND LOCATIONS:
Overall Officials: Inci Yuksek, Study Chair — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus